CLINICAL TRIAL: NCT06028529
Title: Feasibility and Safety of a Portable Exoskeleton to Improve Mobility in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: N4387-P
Record Dates: First submitted 2023-05-30; First posted 2023-09-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease
Keywords: exoskeleton
MeSH Terms: conditions — Parkinson Disease | interventions — Exoskeleton Device

STUDY DESIGN:
Intervention Model Description: Safety, tolerability, feasibility, methodological assessment, and sample characteristics with consideration of multiple staging and high patient variability towards the design of a future clinical efficacy study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Feasibility and Safety (Other): This is a feasibility study to assess the safety and potential utility of a lightweight ground exoskeleton (Keeogo, B-Temia, Inc.) to enhance mobility in people with Parkinson's disease (PD).
  Interventions: Device: Exoskeleton

INTERVENTIONS:
Device: Exoskeleton — lightweight ground exoskeleton
  Other Names: Keeogo

SUMMARY:
Physical therapy approaches for balance and walking deficits in Parkinson's disease (PD) have limited effectiveness, with mostly short-lasting benefits. An exoskeleton is a device that straps to the legs and provides a passive force to assist people to better ambulate. The goal of this study is to establish the feasibility and safety of a lightweight exoskeleton on mobility and fall reduction in people with PD. As most PD patients eventually require assistive mobility devices, the exoskeleton represents a new option for increased, mobility, quality of life, and independence. Qualified subjects will come to the clinic twice weekly for eight weeks (16 total visits) and wear the exoskeleton device while walking under the supervision of a trained kinesiotherapist. Study staff will also interview participants and assess their PD symptoms, quality of life, and overall mobility. This study hopes to establish exoskeletons as modern, standard of care devices, which allow people with PD to maintain more independent and productive lives.

DETAILED DESCRIPTION:
Currently, progressive resistance exercise training, high intensity treadmill training, balanced-based perturbation, and standard physical exercises are utilized to treat mobility deficits associated with PD; however, the effectiveness of these therapies is limited. This study proposes to investigate the utility of a portable exoskeleton for people with PD. The goal is to establish the safety of a lightweight portable exoskeleton, the Keeogo, for gait training and to preliminarily assess its potential efficacy for gait mobility and fall reduction. As the vast majority of PD patients eventually require assistive mobility devices, portable exoskeletons represents an avenue for increased, mobility, quality of life, and independence. Robotic-assist gait training (RAGT) has been extensively applied as a remarkable therapeutic modality, such that it is enabling highly motivated people with devastating neurologic injuries to regain independent ambulation. Despite the potential for this technology to transform the lives of people with PD, these devices are not being adequately investigated in people with movement disorders.

To establish preliminary safety and efficiency of the Keeogo exoskeleton for PD patients at various disease stages, the investigators will examine representative subjects in Hohen & Yahr stages II, III, and IV. Inclusion criteria are: 1) PD confirmed by a PADRECC movement disorder specialist using UK Brain Bank Criteria, 2) Modified H&Y stage II-V. Exclusion criteria are: 1) neurological, musculoskeletal, or other disorders unrelated to PD contributing to impairment of stance, gait, balance or coordination, 2) severe CHF, COPD, or those requiring nasal canula O2, 3) history of implantable cardiac device or ablative surgery, 4) moderate to severe cognitive impairment / dementia (Montreal Cognitive Assessment < 17/30), 5) symptomatic orthostatic hypotension with exertion, 6) feeding tube or associated port placement (PEG/J-PEG), 7) body height less than 5'1" or greater than 6'3" 8) body weight greater than 250 pounds, and 9) amputation of any portion of the lower limbs. Subjects will participate in a total of 30 minutes RAGT ambulation with the Keeogo twice per week for 8 weeks (16 sessions). Subjects may opt to utilize a platform rolling walker, rolling walker, bilateral Lofstrand crutches or a unilateral device, such as a cane or Lofstrand crutch, and will be maintained throughout the intervention.

To establish safety, the number and severity of AEs, such as falls, discomfort, skin or musculoskeletal injury, and orthostatic hypotensive episodes will be documented. Intervention efficacy will be measured pre- and post-donning of the Keeogo exoskeleton at bi-weekly intervention visits, and at 3 post-study visits. Walking capacity, including benefits on FoG, will be assessed with the Six Minute Walk Test (6MWT), balance and postural stability with the MiniBest test, and disease severity with the Examination, Part III, of the Unified Parkinson's Disease Rating Scale (UPDRS). Additional assessments will include surveys about quality of life, activity, balance, and feedback on the device. As a primary end point for establishing efficacy, the 6MWT will be compared between end of training and baseline (with and without the exoskeleton), as well as at 6 and 12 weeks post-study as a durability assessment towards establishing a need for future assessment of in-home usage. These pilot investigations are expected to lay the groundwork for a large multi-center clinical study to establish ground exoskeletons as modern, standard of care devices to aid Veterans and other people with PD and other disabling movement disorders to maintain a more normal and productive life.

ELIGIBILITY:
Inclusion Criteria:

* PD confirmed by a PADRECC movement disorder specialist using UK Brain Bank Criteria
* Modified H&Y stage II-V
* Veteran
* Able to attend visits at the Richmond VA Medical Center

Exclusion Criteria:

* neurological, musculoskeletal, or other disorders unrelated to PD contributing to impairment of stance, gait, balance or coordination
* severe CHF, COPD, or those requiring nasal canula O2
* history of implantable cardiac device or ablative surgery
* moderately-severe to severe cognitive impairment / dementia (Montreal Cognitive Assessment < 17/30)
* symptomatic orthostatic hypotension with exertion
* feeding tube or associated port placement (PEG/J-PEG)
* body height less than 5'1" or greater than 6'3"
* body weight greater than 250 pounds
* amputation of any portion of the lower limbs
* osteoporosis as defined by DEXA Scan T score < -2.5
* failure to meet B-Temia-established hip and knee flexion and extension manual muscle test (MMT) prerequisite screening parameters, which assure that individuals can adequately engage and walk against the resistive forces of the Keeogo
* inability to complete 20 minutes of walking with the exoskeleton (over a maximum period of one hour) at the initial screening/testing session

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Falls While Wearing the Exoskeleton (Safety and Tolerability) Change | Through last training visit (weeks 1-8, 16 sessions)
  Patients will be continuously supervised by a trained physical therapist and the expectation is that there will be no falls while wearing the device. All primary safety and tolerability measures will be separately assessed with consideration of H&Y staging (2-4; max. 5) and cognition (based on MOCA scores 0 = nl, max. 30).
  -Minimal attrition rate based on subjects being unable to complete the protocol. This could for example establish that the Keeogo device is not tolerated by more advanced (H&Y Stage 5) patients, but is acceptable for others.
Incidence of Attrition (Tolerability) Change | Through last training visit (weeks 1-8, 16 sessions)
  The expectation is that there will be minimal attrition rate based on subjects being unable to complete the protocol. In the case of attrition, patients will be interviewed for contributory sources.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) Change | through last training visit (weeks 1-8, 16 sessions)
  Patients will be questioned at the beginning of each session about potential AEs and any AEs observed during sessions by the therapists will be recorded at each training session. The expectation is that there will be no uncorrected and unacceptable AEs as captured by regular structured interviews.
Six-minute Walk Test (Suitability as a Future Primary Efficacy Measure) Change | through last training visit (weeks 1-8, 16 sessions) and 6- and 12-wks post-training
  The suitability of the 6MWT as a future primary clinical outcome measure (and our secondary measures) will be determined from the therapists' impression of ease and reliability of usage and from anticipated trends in scoring improvement. The outcomes here from the 6MWT and secondary measures will be further used towards powering for a future clinical efficacy study, while accounting for preliminary defined influences of severity of PD (H&Y Staging) and cognition (MOCA scoring). Additionally, 6- and 12-weeks post-training assessments will be used to preliminarily assess the durability of training effects.
Patient Satisfaction | immediate post-training
  All subjects will be interviewed for patient satisfaction with wearing and training with the exoskeleton.

SECONDARY OUTCOMES:
Motor examination (Part III) of the modified Unified Parkinson's Disease Rating Scale (Suitability as a Future Secondary Efficacy Measure) | immediate post-training, 6- and 12-wks post-training
  Will assess the suitability of the modified UPDRS Part III (nl = 0, max. 128) as a future secondary clinical outcome measure. Will be collected at baseline and end of training. Additionally, 6- and 12-weeks post-training assessments will be used to preliminarily assess the durability of training effects.
Mini Best Test (Suitability as a Future Secondary Efficacy Measure) | immediate post-training, 6- and 12-wks post-training
  Will assess suitability as a future secondary clinical outcome measure, focused on balance. Additionally, 6- and 12-weeks post-training assessments will be used to preliminarily assess the durability of training effects.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica B Lehosit, Principal Investigator — Richmond VA Medical Center, Richmond, VA
Locations (1):
- Richmond VA Medical Center, Richmond, VA, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No